CLINICAL TRIAL: NCT00884195
Title: Journaling and Weight Loss
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 200816667
Record Dates: First submitted 2009-04-17; First posted 2009-04-20 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Obesity
Keywords: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Gratitude Journaling
  Interventions: Behavioral: Gratitude Journaling
- 2 (Placebo Comparator): Neutral Journaling
  Interventions: Behavioral: Neutral Journaling

INTERVENTIONS:
Behavioral: Gratitude Journaling — Participants will be asked to write down 5 things every day for which they are grateful.
  Arms: 1
Behavioral: Neutral Journaling — Participants will be asked to write down 5 things every day that they noticed about being involved in a weight loss program.
  Arms: 2

SUMMARY:
This is a pilot study to evaluate the effect of keeping a 'gratitude journal' on the outcome of a weight loss program. All the subjects will be enrolled in the Lifesteps weight management program. The experimental group will maintain a gratitude journal and the control group will maintain a 'neutral' journal.

DETAILED DESCRIPTION:
Subjects who are referred to the Preventive Cardiology Program for weight management will be enrolled in the study after obtaining informed consent.

Subjects are enrolled into the program in groups of 10 to 12 every 6 weeks. Alternate groups will be will assigned to the two types of journaling. Each group will be given specific instructions related to the form of journaling assigned. These instructions will be in addition to the usual care prescribed in the Lifesteps® program. In the intervention group, patients will be introduced to gratitude journaling at the beginning of the 12 week class series and asked to journal each day. They will turn in their gratitude journal weekly. At the beginning of each weekly class, five minutes will be spent discussing the journaling.

The control groups will not receive the information on gratitude journaling, but instead will be asked to complete a neutral journal in which they will journal in a general manner regarding their experiences participating in the Lifesteps® weight management program. These will also be collected weekly. At the beginning of class, five minutes will be spent discussing the journaling.

There will be one consent form for the two groups. The instruction (either gratitude journaling or neutral journaling) that will be given to the subjects will reflect the group to which they have been randomized. Both types of journals will be reviewed initially, at mid-point and final by the psychologist (Robert Emmons) to verify the quality of reporting.

Routine tests- Weekly weights

Study Tests:

Pre/post depression: Beck Depression Inventory II; Pre/post Locus of Control: Multidimensional Health Locus of Control Scale; Pre/post SF 36 Quality of Life Questionnaire; Pre/post Gratitude Questionnaire

ELIGIBILITY:
Inclusion Criteria:

* BMI>25
* >18 years of age

Exclusion Criteria:

* Severe psychiatric diagnosis which in the opinion of the PI would compromise participation in the study.
* Addiction to alcohol and drugs

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-01 (Actual); Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Weight loss | 3 months

SECONDARY OUTCOMES:
Quality of Life | 3 months
Class attendance | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: CT Kappagoda, MD, PhD, Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis Medical Center, Sacramento, California, United States